CLINICAL TRIAL: NCT05067244
Title: A Phase 2 Open-Label Treatment Development Study of MDMA-Assisted Cognitive Processing Therapy (CPT) for Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Remedy (Industry)
Collaborators: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-087
Record Dates: First submitted 2021-09-19; First posted 2021-10-05 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: MDMA; Cognitive Processing Therapy (CPT)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MDMA assisted psychotherapy (Experimental): Participants will undergo a 2-month course of CPT psychotherapy for PTSD with two sessions that integrate MDMA-assisted psychotherapy. MDMA will be administered ini two separate sessions and integrated into the psychotherapy protocol. The two doses of MDMA during this study will be used as an adjunct to psychotherapy.
  Interventions: Drug: MDMA

INTERVENTIONS:
Drug: MDMA — MDMA assisted psychotherapy

SUMMARY:
This study is designed to provide information on whether the drug MDMA, combined with Cognitive Processing Therapy (CPT), is safe and helpful for people with Post Traumatic Stress Disorder (PTSD). PTSD is a serious debilitating disorder that negatively impacts a person's daily life, and can result in diminished functioning, fractured relationships, inability to maintain employment, substance abuse, depression, and suicide risk. People who suffer from PTSD relive their traumatic experience(s) through nightmares and flashbacks, have difficulty sleeping, and feel detached or estranged.

CPT is a manualized treatment for PTSD, which has the participant make meaning of the traumatic event and its impact on their life. CPT is one of the treatments with the best evidence for the treatment of PTSD to date. Clients with PTSD discuss how they believe the trauma has impacted them, and the therapist teaches the client skills to challenge areas where they are "stuck" remembering the traumatic event.

MDMA is a drug commonly used recreationally that has been increasingly studied because of its ability to reduce the impact of PTSD symptoms. The effects of MDMA are reduced fear, enhanced communication, trust and introspection, and increased empathy and compassion. The effects of MDMA create a state that enhances the positive effects of therapy by increasing the ability to tolerate negative emotions and allowing clients to stay engaged in therapy without being overwhelmed by the intense emotions surrounding the memories of traumatic events. It is believed that MDMA may help promote the effects of CPT. Given the properties of MDMA, specifically in inducing the ability to stay with emotion and challenging cognitions, these effects are especially relevant to the mechanisms of CPT.

This is a pilot study exploring CPT integrated with MDMA-assisted psychotherapy for treatment of PTSD. This study will enroll 10 participants diagnosed with PTSD, who will undergo a 2-month course of psychotherapy that includes CPT integrated with MDMA-assisted psychotherapy. Participants will go through CPT sessions, and two doses of MDMA will be used as an adjunct to psychotherapy. Since this is the first time that CPT is being combined with individual MDMA-assisted psychotherapy for PTSD, the researchers are interested in gathering preliminary information about the blending of these two therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Meet criteria for PTSD
2. Are at least 18 years old
3. Are a resident of Ontario and live within 200km of the study site
4. Are in good physical health
5. Are proficient in speaking and reading English
6. Are willing to have all visits audio and video recorded
7. Are able to swallow pills
8. Agree to all study rules and commit to all medical and therapy visits
9. If in psychotherapy, are willing to allow the study therapists to communicate directly with your therapist
10. Are willing to stop taking psychiatric medications, herbal supplements, prescription and nonprescription medications during the study
11. Agree not to drive for at least 24 hours after taking MDMA
12. Agree to stay overnight on two separate occasions after each full-day MDMA-Assisted Psychotherapy Session
13. Are not pregnant and will commit to not becoming pregnant during the study, if you are able to become pregnant
14. Have a supportive relative, spouse, close friend or other caregiver who can serve as your emergency contact
15. Agree to inform the researchers within 48 hours of any medical conditions and procedures
16. Agree to not participate in any other clinical trials during this study

Exclusion Criteria:

1. Are pregnant or could become pregnant and not using birth control
2. Have a history of, or a current psychotic disorder, bipolar 1 disorder or dissociative identity disorder
3. Have a history of a medical condition that could make receiving MDMA unsafe (e.g. glaucoma, heart attack, stroke, aneurysm)
4. Have a history of Diabetes Mellitus (Type 2) that a doctor determines is not stable
5. Have hypothyroidism (low activity in the thyroid gland) and are not on thyroid replacement
6. Have high blood pressure, a history of heart disease, heart failure, irregular activity in the heart or require heart medication
7. Have liver disease with symptoms
8. Have history of hyponatremia (when you have decreased levels of sodium in the blood, which can cause confusion, seizures, fatigue and low levels of consciousness)
9. Have history of hyperthermia (when you have a dangerously overheated body, usually in response to hot, humid weather)
10. Weigh less than 48 kg
11. Have recently engaged in suicidal behavior or had serious suicidal thoughts (this will be assessed by a therapist)
12. Require ongoing therapy with a psychiatric medication
13. Have a current eating disorder with active purging
14. Have current major depressive disorder with psychotic features
15. Are a serious risk to others
16. Have recently received Electroconvulsive Therapy (ECT)
17. Have recently engaged in ketamine-assisted therapy or used ketamine
18. Have current substance use disorder (not including caffeine or nicotine)
19. Have recently used "Ecstasy" (material represented as containing MDMA)
20. Are not able to give adequate informed consent
21. Are not able to adhere to the requirements for procedures, attendance and timing of visits, and observe limits regarding study staff time and support as indicated by a time-limited clinical trial
22. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline to Primary Endpoint in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Score | Baseline (enrolment) to endpoint (6 month follow up)
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Change From Baseline to Midpoint (visit 6) in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Score | Baseline (enrolment) to midpoint (visit 6, 3-4 weeks)
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Change From Baseline to 1 Month Follow up in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Score | Baseline (enrolment) to 1 month follow up
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Change From Baseline to 3 Month Follow up in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Score | Baseline (enrolment) to 3 month follow up
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.

SECONDARY OUTCOMES:
Change From Baseline to Endpoint in PTSD Symptoms Checklist | Baseline (enrolment) to endpoint (6 month follow up)
  PTSD Checklist for the DSM-5 (PCL-5) is a self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the DSM-5 symptoms of PTSD. Participants indicate how much distress they have experienced due to symptoms on a five-point Likert-type scale (1 = not at all, 5 = extremely). The total PCL-5 score (a sum of all 20 items) provides an index of overall PTSD symptom severity with higher scores indicating higher severity.
Change From Baseline to Midpoint (Visit 6) in PTSD Symptoms Checklist | Baseline (enrolment) to midpoint (visit 6, 3-4 weeks)
  PTSD Checklist for the DSM-5 (PCL-5) is a self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the DSM-5 symptoms of PTSD. Participants indicate how much distress they have experienced due to symptoms on a five-point Likert-type scale (1 = not at all, 5 = extremely). The total PCL-5 score (a sum of all 20 items) provides an index of overall PTSD symptom severity with higher scores indicating higher severity.
Change From Baseline to 1 Month Follow up in PTSD Symptoms Checklist | Baseline (enrolment) to 1 month follow up
  PTSD Checklist for the DSM-5 (PCL-5) is a self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the DSM-5 symptoms of PTSD. Participants indicate how much distress they have experienced due to symptoms on a five-point Likert-type scale (1 = not at all, 5 = extremely). The total PCL-5 score (a sum of all 20 items) provides an index of overall PTSD symptom severity with higher scores indicating higher severity.
Change From Baseline to 3 Month Follow up in PTSD Symptoms Checklist | Baseline (enrolment) to 3 month follow up
  PTSD Checklist for the DSM-5 (PCL-5) is a self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the DSM-5 symptoms of PTSD. Participants indicate how much distress they have experienced due to symptoms on a five-point Likert-type scale (1 = not at all, 5 = extremely). The total PCL-5 score (a sum of all 20 items) provides an index of overall PTSD symptom severity with higher scores indicating higher severity.
Change From Baseline to Endpoint in The Patient Health Questionnaire-9 Depression Symptoms | Baseline (enrolment) to endpoint (6 month follow up)
  The Patient Health Questionnaire-9 (PHQ-9) is used to assess depressive symptom severity. The PHQ-9 includes items which correspond with the diagnostic criteria for DSM-IV major depressive disorder. Scores can indicate either no depression, minimal, mild, moderate, moderately severe, or severe depression. Higher scores indicate higher severity in depressive symptoms.
Change From Baseline to Midpoint (Visit 6) in The Patient Health Questionnaire-9 Depression Symptoms | Baseline (enrolment) to midpoint (visit 6, 3-4 weeks)
  The Patient Health Questionnaire-9 (PHQ-9) is used to assess depressive symptom severity. The PHQ-9 includes items which correspond with the diagnostic criteria for DSM-IV major depressive disorder. Scores can indicate either no depression, minimal, mild, moderate, moderately severe, or severe depression. Higher scores indicate higher severity in depressive symptoms.
Change From Baseline to 1 Month Follow up in The Patient Health Questionnaire-9 Depression Symptoms | Baseline (enrolment) to 1 month follow up
  The Patient Health Questionnaire-9 (PHQ-9) is used to assess depressive symptom severity. The PHQ-9 includes items which correspond with the diagnostic criteria for DSM-IV major depressive disorder. Scores can indicate either no depression, minimal, mild, moderate, moderately severe, or severe depression. Higher scores indicate higher severity in depressive symptoms.
Change From Baseline to 3 Month Follow up in The Patient Health Questionnaire-9 Depression Symptoms | Baseline (enrolment) to 3 month follow up
  The Patient Health Questionnaire-9 (PHQ-9) is used to assess depressive symptom severity. The PHQ-9 includes items which correspond with the diagnostic criteria for DSM-IV major depressive disorder. Scores can indicate either no depression, minimal, mild, moderate, moderately severe, or severe depression. Higher scores indicate higher severity in depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Bruni, MD, Principal Investigator — Remedy Institute; Anne Wagner, PhD, Study Chair — Remedy Institute
Locations (1):
- Remedy Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No